CLINICAL TRIAL: NCT02131090
Title: A Comparison of Intrapartum Epidural Fixation Devices: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Epi devices RCT
Record Dates: First submitted 2014-03-31; First posted 2014-05-06 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Labour; Childbirth
Keywords: Epidural; Catheter; Fixation; Device; Intrapartum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tegaderm TM (Experimental): Participants in this arm of the study will receive the Tegaderm dressing to secure the epidural catheter
  Interventions: Device: Tegaderm TM
- Lock-it Plus (Experimental): Participants in this arm of the study will receive the Lock-it Plus dressing to secure the epidural catheter
  Interventions: Device: Lock-it Plus
- Epifix (Experimental): Participants in this arm of the study will receive the Epifix dressing to secure the epidural catheter
  Interventions: Device: Epifix

INTERVENTIONS:
Device: Tegaderm TM — This is a generic adhesive dressing which is commonly used to secure epidural catheters.
  Arms: Tegaderm TM
Device: Lock-it Plus — This dressing is specifically designed for securing epidural catheters. It is adhesive to the patient's back and has a plastic clamp through which the epidural catheter passes. Once closed, the clamp secures the catheter.
  Other Names: Manufactured by Smith's Medical
  Arms: Lock-it Plus
Device: Epifix — This dressing is specifically designed to secure epidural catheters. It is adhesive to the patient's back and has a foam, moulded mechanism through which the catheter is passed. An adhesive flap folds over the whole mechanism to secure the catheter.
  Other Names: Epifix is manufactured by Unomedical
  Arms: Epifix

SUMMARY:
A number of methods are currently used to prevent movement of epidural catheters in women during labour. These usually consist of sticky dressings applied to the patient's back. The purpose of this study is to compare how much epidural catheters move when secured with three commonly used different fixation dressings with the aim of identifying the best method of securing epidural catheters.

Movement of epidural catheters has several clinical implications. Usually only a short length of epidural catheter is left in the epidural space, and therefore any significant movement could result in the catheter moving out of the epidural space leading to a loss of the pain relieving effects of the epidural.

Once epidural failure has occurred due to catheter migration, a second catheter must be inserted in order to re-establish pain relief and thus the patient is exposed to the risks of epidural insertion for a second time.

If the researchers in this study can identify a method of fixing epidural catheters which results in the least amount of catheter movement, then patients could benefit from more reliable epidural pain relief, fewer repeated procedures and the risks associated with repeated procedures.

The principle objective of the study is to determine which epidural fixation dressing results in the least amount of epidural catheter movement from the time of epidural insertion (during labour) to the time of epidural removal (after labour).

DETAILED DESCRIPTION:
The null hypothesis is that there is no difference in epidural catheter migration between any of the epidural catheter fixation devices.

The study design has been chosen so that the researchers can fairly assess how different commercially available epidural fixation devices perform in the real life scenario of labour, a time when epidurals are particularly important to the well-being of a labouring woman. Three different epidural fixation methods will be studied. These three methods have been chosen because they are all already in use in different hospitals across the UK but have never been compared together.

1. Women admitted to labour ward at St. George's Hospital will be invited to participate in the study. Written informed consent will be obtained from all potential participants.
2. Women in labour who request an epidural will be randomly allocated to one of three different dressings used to secure the epidural. The epidural will be performed by the duty anaesthetist according to a standard practice. The three epidural dressings are: 3M Tegaderm, Smiths Medical Lockit Plus and Unomedical Epifix. All dressing will be applied in a standardised manner. Since 3M Tegaderm is the current dressing used at St. George's Hospital it will form the control group.
3. Epidurals will be inserted by the duty anaesthetist using a standard technique and the appropriate dressing applied. In order to avoid bias women will not be informed which device they are to receive.
4. Patient characteristics will be documented for each epidural, including length of catheter at skin at time of insertion, depth to epidural space, intervertebral interspace used (e.g. L3-4), patient position for epidural insertion (lateral or sitting), time and date of epidural insertion, patient body mass index (at booking). No identifying patient data will be recorded.
5. If an epidural is removed before delivery or the epidural fixation device is altered then the reason for intervention will be documented e.g. inadequacy of epidural analgesia, loss of integrity of fixation device. Any specific events that precipitate problems with the epidural fixation devices will be documented e.g. discomfort at site of dressing on transfer of patient onto operating theatre table.
6. After delivery of the baby, the epidural catheter will be removed. Removal will be encouraged within the first hour following delivery and before the patient has mobilised from their bed. If possible then the woman will adopt the same position (either sitting or lateral) for removal of the epidural as she was in for insertion. Removal of the catheter will either be by a midwife or the duty anaesthetist.
7. After removal of the epidural the following patient characteristics will be collected by the midwife or anaesthetist removing the catheter: length of catheter at skin at time of removal, patient position for epidural removal (lateral or sitting), time and date of epidural removal, integrity of epidural dressing, whether the patient was transferred to the operating theatre table, any additional problems encountered with the epidural or dressing.
8. No specific restrictions will be placed on participants following epidural insertion, other than those that are routine for all labouring women with epidurals. However any women who move off their bed and walk before removal of their epidural catheter will be excluded from the study, since walking may cause the epidural catheter to migrate more than it would do so usually during labour.

Data will be analysed to determine whether the null hypothesis is accepted or rejected. Information about the study and any conclusion drawn will be published locally and nationally in order to inform decision making regarding which epidural catheter fixation device is best suited to reduce epidural migration in labouring women.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Patient in labour, requesting an epidural.
* Primi-parous women
* Multi-parous women
* BMI < 50

Exclusion Criteria:

* BMI >50
* Documented diagnosis of scoliosis and/or other significant lumbar spinal pathology
* Previous lumbar spinal surgery
* Any contraindication to epidural analgesia
* Unable to consent for inclusion in study
* Admitted for termination of pregnancy or intra-uterine death

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Migration of epidural catheter in centimetres | Upon epidural removal within 1 hour from delivery

SECONDARY OUTCOMES:
Comfort of each fixation device for women during labour. | Upon epidural removal within 1 hour from delivery
  A simple questionnaire incorporated into the data collection sheet, section 3. Women will be asked whether the dressing was comfortable and their response will be recorded as either 'comfortable' or 'uncomfortable'
Structural integrity of each dressing. | Upon epidural removal within 1 hour from delivery
  This will be assessed using a simple questionnaire as part of the data collection form in section 2. The midwife removing the epidural will record whether the dressing is either 'intact', 'partially peeled off' or 'completely peeled off'.
Rate of epidural failures associated with each fixation device. | Upon epidural removal within 1 hour from delivery
  Assessed using the data collection questionnaire section 3. Data collectors will answer two questions:
  Has the epidural block partially failed? Yes or No.
  Partial failure is defined as pain despite epidural top ups, but not requiring the epidural to be re-sited.
  Has the epidural block completely failed? Yes or no.
  An epidural is defined as 'completely failed' if it needs to be re-sited at any point during labour.
Effect of Body Mass Index on dressing integrity | Upon epidural removal within 1 hour from delivery
  The Body Mass Index (BMI) of each participant will be recorded. This data will be correlated with each dressing type and data collected regarding device integrity as collected in the data collection form section 2 as previously described.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Odor, Study Chair — St George's, University of London; sohail Bampoe, Principal Investigator — St George's, University of London
Locations (1):
- St. Georges Hospital NHS Trust, London, Tooting, United Kingdom